CLINICAL TRIAL: NCT06063980
Title: Sinus Augmentation in the Posterior Maxillary Region: a Case Report of 0mm Bone
Brief Title: Sinus Augmentation in the Posterior Maxillary Region: a Case Report of 0mm Bone Height.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VNU University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Pham Nhu Hai, Associate professor, VNU University of Medicine and Pharmacy
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VNUMed
Record Dates: First submitted 2023-09-19; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Bone Resorption
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional sinus lift procedure (Other): Participants assigned to conventional sinus augmentation
  Interventions: Procedure: Conventional sinus lift surgery
- Two-stage-sinus-lift procedure (Other): Participants assigned to two-stage - sinus - lift procedure
  Interventions: Procedure: Two-stage-sinus-lift procedure

INTERVENTIONS:
Procedure: Conventional sinus lift surgery — After graft reflection, sinus membrane is separated from bone or oral mucosa and then bone graft is inserted in between the two structures.
  Arms: Conventional sinus lift procedure
Procedure: Two-stage-sinus-lift procedure — Procedure is performed in two stages with the purpose of stage one to separate the oral mucosa from the sinus membrane using a small amount of bone graft and stage two as actual sinus augmentation, which is performed similar to that of conventional sinus lift procedure.
  Arms: Two-stage-sinus-lift procedure

SUMMARY:
Sinus floor elevation (SFA) and GBR have been applied in the placement of dental implants in longstanding edentate posterior maxilla region. However, the number of study on the efficacy of these procedure on areas with 0mm bone height is limited. This case study aims to compare two cases of 0mm bone height in the posterior maxillae region with different handling procedure. In this article, two female patients in their 40s underwent maxillary sinus augmentation (sinus lifting) due to longstanding missing posterior maxillary molars with the bone of which area had resorbed entirely, leaving 0mm bone height. One patient went through conventional sinus augmentation while the other had a two-stage - sinus - lift procedure. Researchers compared the bone - volume induced between the two procedures.

ELIGIBILITY:
Inclusion Criteria:

* 0mm bone height at posterior maxillae region

Exclusion Criteria:

* general contraindication to implant surgery
* subjected to irradiation in the head and neck area <1 one year before implantation
* uncontrolled diabetes
* pregnant or nursing
* substance abuse
* heavy smoker
* psychiatric therapy or unrealistic expectations
* immunosuppressed or immunocompromised
* treated or under treatment with oral or intravenous aminobisphosphonates
* untreated periodontitis
* poor oral hygiene and motivation

Ages: 40 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2021-09-25 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Bone formation recorded after two-step-sinus-augmentation. | 21 months
  9,98mm bone height is recorded on CBCT.

CONTACTS AND LOCATIONS:
Locations (1):
- VNU University of Medicine and Pharmacy, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided